CLINICAL TRIAL: NCT03498313
Title: Unique Effects of Perimenstrual Estradiol or Progesterone Supplementation on Perimenstrual Suicidality
Acronym: CLEAR-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tory Anne Eisenlohr-Moul, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-0189; R00MH109667 (NIH)
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Suicidal Ideation
Keywords: steroid hormones; estradiol; estrogen; progesterone; depression; suicide
MeSH Terms: conditions — Suicidal Ideation; Depression; Suicide | interventions — Estradiol; Sugars; Progesterone

STUDY DESIGN:
Intervention Model Description: Crossover 3-condition placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Transdermal Estradiol + Placebo (Experimental): .1mg per 24 hours transdermal estradiol applied to the skin weekly, and sugar pill manufactured to mimic the progesterone pills taken twice daily by mouth, for 14 days.
  Interventions: Drug: Transdermal Estradiol + Placebo
- Oral Micronized Progesterone + Placebo (Experimental): 100 mg oral micronized progesterone pill taken twice daily by mouth, and clear patch manufactured to mimic the E2 patch applied to the skin weekly, for 14 days.
  Interventions: Drug: Oral Micronized Progesterone + Placebo
- Placebos (Placebo Comparator): Sugar pill designed to mimic the P4 pills taken twice daily by mouth, and clear patch manufactured to mimic the E2 patch applied to the skin weekly, for 14 days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Transdermal Estradiol + Placebo — .1mg/24hr transdermal estradiol for 14 days starting day 7 after positive urine luteinizing hormone test, plus twice daily placebo pills during the same time frame.
  Other Names: Climara; sugar pill
  Arms: Transdermal Estradiol + Placebo
Drug: Oral Micronized Progesterone + Placebo — 100mg oral micronized progesterone twice daily for 14 days starting day 7 after positive urine luteinizing hormone test, plus weekly application of a placebo patch during the same time frame.
  Other Names: Prometrium; placebo patch
  Arms: Oral Micronized Progesterone + Placebo
Drug: Placebos — Twice daily placebo pills for 14 days starting day 7 after positive urine luteinizing hormone test, plus weekly application of a placebo patch during the same time frame.
  Other Names: sugar pill; placebo patch
  Arms: Placebos

SUMMARY:
This within-person, crossover, 3-condition, placebo-controlled study compares the impact of three perimenstrual conditions on severity of suicidal symptoms in females with past-month suicidality but minimal risk of imminent suicide attempt. The three conditions are (1) perimenstrual withdrawal from estradiol only (during progesterone stabilization), (2) perimenstrual withdrawal from progesterone only (during estradiol stabilization), and (3) perimenstrual withdrawal from both estradiol and progesterone during placebo.

DETAILED DESCRIPTION:
Previous work from our group demonstrates that perimenstrual worsening of suicidal thoughts in females is caused by normal perimenstrual withdrawal from the ovarian steroids estradiol (E2) and progesterone (P4), since perimenstrual stabilization of E2+P4 prevented the perimenstrual worsening of suicidal ideation observed under placebo. In the present study, we follow up on that work with an additional mechanistic trial in which E2 and P4 will be stabilized in separate arms of the study.

60 (30 completers) female outpatients, with past-month suicidal ideation but minimal imminent risk for attempt, will complete self-reports and clinical interviews measuring presence and severity of suicidal ideation in each of three conditions (A, B, C: order randomized across three menstrual cycles): (A) perimenstrual E2/P4 withdrawal (under placebo), (B) perimenstrual P4 withdrawal (exogenous stabilization of E2 only), and (C) perimenstrual E2 withdrawal (exogenous stabilization of P4 only). A washout cycle will separate conditions. Analyses will compare the perimenstrual trajectories of symptoms and suicidality across the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adhere to medication regimen
* Speaks English
* Assigned female at birth with intact ovaries
* Premenopausal
* Normal menstrual cycles between 25-35 days
* Under current care of an outpatient mental health provider with visits occurring at least once every 3 months.
* At least 1 year postpartum.
* Willing to use a barrier method of birth control during the study.
* Normal weight (BMI between 18.00-29.99)
* Must report at least some recent suicidal ideation (in the past month) at the time of recruitment.
* Must be categorized as having acceptably low imminent risk for suicidal crisis/attempt by a licensed clinical psychologist utilizing evidence-based clinical and research guidelines for imminent suicide risk management.

Exclusion Criteria:

* Must not be pregnant, breastfeeding, or trying to become pregnant.
* Must not be taking any form of exogenous hormones or hormonal intrauterine device, and must have ended previous use of hormonal preparations at least one month prior to the study.
* Must not have a personal history of any chronic medical condition that may interfere with the aims of the study or make the experimental protocol unsafe, including but not limited to metabolic or autoimmune disease, epilepsy, endometriosis, cancer, diabetes, cardiovascular, gastrointestinal, hepatic, renal, or pulmonary disease, and no personal or first degree family history of thromboembolic events.
* Any current cigarette smoking is exclusionary.
* Must not report a current diagnosis of major depressive episode with peripartum onset (current episode), and must not be currently receiving treatment for premenstrual dysphoric disorder (Note: Premenstrual Dysphoric Disorder diagnosis must have been made based on prospective daily ratings).
* Must not report any history of manic episode, any history of psychotic symptoms, or current substance use disorder.
* Must not test positive for (unprescribed) opioid use, methamphetamine use, or cocaine use at the start of an experimental condition.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tory A Eisenlohr-Moul, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Neuropsychiatric Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were enrolled (consented) in the study. Following a baseline phase in which participants completed daily symptom ratings and prepared to begin urinary LH testing as part of the lead-up to the first experimental period, 46 participants remained in the study and were randomized to one of six sequences of the three experimental conditions.
Groups:
- E-P-PBO: Estrogen First, then Progesterone, then Placebo
- E-PBO-P: Estrogen, Placebo, Progesterone
- P-E-PBO: Progesterone, Estrogen, Placebo
- P-PBO-E: Progesterone, Placebo, Estrogen
- PBO-E-P: Placebo, Estrogen, Progesterone
- PBO-P-E: Placebo, Progesterone, Estrogen
Period: Experimental Period 1
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E
Started | 9 | 8 | 9 | 5 | 9 | 6
Completed | 8 | 7 | 9 | 4 | 9 | 6
Not Completed | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E
Started | 8 | 7 | 9 | 4 | 9 | 6
Completed | 7 | 4 | 9 | 3 | 9 | 5
Not Completed | 1 | 3 | 0 | 1 | 0 | 1
Not completed — Anovulation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1 | 0 | 1
Period: Experimental Period 2
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E
Started | 7 | 4 | 9 | 3 | 9 | 5
Completed | 7 | 4 | 9 | 3 | 8 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2
Period: Washout Period 2
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E
Started | 7 | 4 | 9 | 3 | 8 | 3
Completed | 3 | 2 | 9 | 2 | 6 | 1
Not Completed | 4 | 2 | 0 | 1 | 2 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0 | 2 | 0
Not completed — Anovulation | 0 | 0 | 0 | 0 | 0 | 1
Period: Experimental Period 3
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E
Started | 3 | 2 | 9 | 2 | 6 | 1
Completed | 3 | 2 | 9 | 2 | 6 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-P-PBO | E-PBO-P | P-E-PBO | P-PBO-E | PBO-E-P | PBO-P-E | Total
Number analyzed (Participants) | 9 | 8 | 9 | 5 | 9 | 6 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 9 | 5 | 9 | 6 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 5 | 9 | 6 | 46
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 1 | 0 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 4 | 0 | 2 | 2 | 8
  White | 6 | 6 | 4 | 4 | 6 | 1 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 9 | 5 | 9 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: Cyclical Change in Suicidal Ideation (SI) Severity
Description: Each day, participants completed five items from the Adult Suicidal Ideation Questionnaire (ASIQ; items 1,2,9,17,19). Response options ranged from 1 (no suicidal ideation) to 6 (extreme severity of suicidal ideation). For each participant on each day, "mean daily SI" was calculated as the mean of these five items.
  Our outcome, Cyclical Change in SI Severity, is calculated for each person, in each condition, as the DIFFERENCE between mean daily SI during the low-risk early luteal phase days (days LH surge +1,2,3,4,5,6,7) and the high-risk perimenstrual phase days (days LH surge +11,12,13,14,15,16,17), with the subtraction carried out as Perimenstrual mean minus Early Luteal mean. Therefore, this single value represents the degree to which an individual showed perimenstrual worsening of SI within a condition.
Time Frame: Days 1 to 17 following positive LH test
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Transdermal Estradiol + Placebo | Oral Micronized Progesterone + Placebo | Placebos
Number analyzed (Participants) | 38 | 35 | 35
units on a scale | -.22 (.05) | -.05 (.07) | .25 (.11)
Statistical Analysis 1: Comparison: Transdermal Estradiol + Placebo vs Placebos; Fixed interaction effect of treatment (0=Placebo, 1=E2) by cycle phase (0=Lower-Risk Early Luteal Baseline, 1=Higher-Risk Perimenstrual Phase) predicting SI severity in a multilevel model (with daily observations nested within conditions nested within participants over time); Test type: Superiority; p = .002, Mixed Models Analysis; This is the p-value for the Treatment X Cycle Phase Interaction. Kenward-Roger Method was utilized for degrees of freedom; Slope = -.25, 95% CI 2-sided [-.41 to -.08], Standard Error of Mean .082 — Placebo represents the reference treatment
Statistical Analysis 2: Comparison: Oral Micronized Progesterone + Placebo vs Placebos; Fixed interaction effect of treatment (0=Placebo, 1=P4) by cycle phase (0=Lower-Risk Early Luteal Baseline, 1=Higher-Risk Perimenstrual Phase) predicting SI severity in a multilevel model (with daily observations nested within conditions nested within participants over time); Test type: Superiority; p = .46, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -.06, 95% CI 2-sided [-.22 to .10], Standard Error of Mean .083 — Placebo Represents the Reference Condition

ADVERSE EVENTS:
Time Frame: Three different two-week conditions, each with at least one month washout between (i.e., 6 weeks total).
Description: Adverse events were assessed via phone daily during the six weeks of medication use.
Arm/Group | Transdermal Estradiol + Placebo | Oral Micronized Progesterone + Placebo | Placebos
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 2/35 | 0/35
Other Adverse Events (participants affected / at risk) | 15/38 | 10/35 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol + Placebo (N=38) | Oral Micronized Progesterone + Placebo (N=35) | Placebos (N=35)
Hospitalization for Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization for Worsening Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol + Placebo (N=38) | Oral Micronized Progesterone + Placebo (N=35) | Placebos (N=35)
Headache (General disorders) | 4 (4) | 5 (5) | 6 (6)
Breast Discomfort (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 4 (4)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (General disorders) | 2 (2) | 2 (2) | 3 (3)
Skin Irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Changes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Self-Report of Adverse Mood Changes (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03498313/Prot_SAP_000.pdf